CLINICAL TRIAL: NCT00322426
Title: Effect of Randomized Patient-Triggered Sensory Cues for Freezing of Gait in Parkinson's Disease
Brief Title: Sensory Cues for Freezing in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Austin Health (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1-Schoffer
Record Dates: First submitted 2006-05-03; First posted 2006-05-05 (Estimated); Last update posted 2006-06-23 (Estimated); Status verified 2006-05

CONDITIONS: Parkinson's Disease
Keywords: Freezing of Gait; Parkinson's Disease; Sensory Cues
MeSH Terms: conditions — Parkinson Disease

INTERVENTIONS:
Device: Sensory Cueing Device

SUMMARY:
The purpose of this study is (1) to determine if patient triggered sensory(auditory, visual and tactile) cues can help treat freezing of gait in Parkinson's disease, and (2) to assess if unexpected (randomized) cues are more effective than anticipated ones.

DETAILED DESCRIPTION:
Freezing of gait (FOG) is defined as a transient halt in motor activity, wherein the patient appears "as if nailed to the floor." It is a common phenomenon in Parkinson's disease (PD), both when medications are at their peak ("on state") and at their lowest effectiveness ("off state"). While "off" FOG often responds to dopaminergic medications, "on" FOG is a difficult to treat, causing significant distress for the patient, and elevating risk of falls and morbidity.

A few small studies have suggested that auditory and visual sensory cues, in the form of continuous stimuli such as a clicking metronome, music, or horizontal lines drawn the floor, may help patients with gait freezing. In this study, we aim to: (1) evaluate if stimuli (including visual, auditory as well as tactile cues) which are present only on patient triggering are effective for FOG in PD; (2) investigate if presentation of unexpected cues, in the form of randomized sensory stimuli, are more effective that anticipated cues.

Participants will include patients diagnosed with PD, stabilized on drug therapy, with adequate vision, hearing, and mentation to respond to cuing, and experiencing "on" FOG. Patients will be evaluated during a single session. A small device which we have developed will be placed around the neck, and emit either repetitive beeping, a flashing line on the floor, or a slight vibration felt over the neck when the patient presses a button on the front panel in response to FOG. Participants will be videotaped walking a 15 m strip with: (1) no cues; (2) auditory cues only; (3) visual cues only; (4) tactile cues only; and (5) randomized cues. The order in which patients receive the cues will be randomized.

A reviewer will watch the videotape with sound off so that they will be blinded to the cues. The Total Time, Freezing Time (duration of walk in which patient experiences freezing, Walking Time (duration of walk during which patient is not experiencing freezing), and Average Duration of Freeze will be recorded for each walk.

ELIGIBILITY:
Inclusion Criteria:

* Currently living in Melbourne, Australia (note that we cannot respond to enquiries from outside of this area)
* Confirmed diagnosis of Parkinson's disease
* Stabilized drug therapy for at least 1 month prior to the study and during
* Hearing and vision - Able to identify lines on floor, hear metronome
* MMSE >24
* Able to walk independently (with or without a mechanical aid)
* Able to give informed consent

Exclusion Criteria:

* Severe comorbidity (joint problems, neuromuscular disorder affecting mobility)
* Severe dyskinesias

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-07; Study Completion 2007-01

PRIMARY OUTCOMES:
Total walking time
Number of freezes
Freeze time - duration of walk in which patient experiences freezing
Walking time - duration of walk during which patient is not experiencing freezing
Average duration of freeze

CONTACTS AND LOCATIONS:
Overall Officials: Kerrie Schoffer, MD, Principal Investigator — Austin Hospital, Melbourne Australia
Locations (1):
- Austin Hospital, Melbourne, Victoria, Australia